CLINICAL TRIAL: NCT00001288
Title: Cerebral Blood Flow Studies of Language and Memory
Brief Title: Brain Blood Flow Studies of Language and Memory
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 910134; 91-N-0134
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-06

CONDITIONS: Cerebrovascular Disorder; Epilepsy
Keywords: Positron Emission Tomography; Epilepsy; Stroke
MeSH Terms: conditions — Cerebrovascular Disorders; Epilepsy; Stroke

INTERVENTIONS:
Drug: 15 O Water
Drug: FDG

SUMMARY:
Positron Emission Tomography (PET) is a technique used to investigate the functional activity of the brain. The PET technique allows doctors to study the normal processes of the brain (central nervous system) of normal individuals and patients with neurologic illnesses without physical / structural damage to the brain.

When a region of the brain is active, it uses more fuel in the form of oxygen and sugar (glucose). As the brain uses more fuel it produces more waste products, carbon dioxide and water. Blood carries fuel to the brain and waste products away from the brain. As brain activity increases blood flow to and from the area of activity increases also. Knowing these facts, researchers can use radioactive water (H215O) and PET scans to observe what areas of the brain are receiving more blood flow.

This study is designed to use positron emission tomography (PET) with radioactive water (H215O) to determine the areas of the brain associated with memory and language. Patients participating in the study will be made up of normal volunteers, patients with epilepsy, and patients with other abnormalities related to the surface of the brain (non-epileptic focal cortical dysfunctions).

DETAILED DESCRIPTION:
This protocol will use positron emission tomography (PET) with H2015 and functional MRI to examine localization of memory and language in normal control subjects, and patients with localization-related epilepsy.

ELIGIBILITY:
INCLUSION CRITERIA:

Normal Volunteers:

The desired age range is 18 to 55 years.

Subjects will have no history of head injury or other neurological disease and must not be taking any medication.

Female subjects of childbearing potential will be administered a pregnancy test; these subjects will not be eligible for the study requiring 2 scans.

All volunteers will read and sign the consent form.

Patients:

Patients will be selected from among those referred to the Clinical Epilepsy Section, NINDS for evaluation.

EXCLUSION CRITERIA:

Patients with evidence of a progressive intracranial process, who are taking any drugs (except AEDs) that might affect the results, or active systemic disease will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 303
Dates: Start 1991-05; Study Completion 2003-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Albert MS, Butters N, Brandt J. Memory for remote events in alcoholics. J Stud Alcohol. 1980 Nov;41(11):1071-81. doi: 10.15288/jsa.1980.41.1071. No abstract available. PMID 7278254
- [Background] Milner B. Interhemispheric differences in the localization of psychological processes in man. Br Med Bull. 1971 Sep;27(3):272-7. doi: 10.1093/oxfordjournals.bmb.a070866. No abstract available. PMID 4937273
- [Background] Petersen SE, Fox PT, Posner MI, Mintun M, Raichle ME. Positron emission tomographic studies of the cortical anatomy of single-word processing. Nature. 1988 Feb 18;331(6157):585-9. doi: 10.1038/331585a0. PMID 3277066